CLINICAL TRIAL: NCT05357898
Title: A Phase 1/2, First-in-Human, Multicenter, Open-Label Study of SQZ-eAPC-HPV as Monotherapy and in Combination With Immune Checkpoint Inhibitor(s) in Patients With HPV16+ Recurrent, Locally Advanced, or Metastatic Solid Tumors
Brief Title: Study of SQZ-eAPC-HPV in Patients With HPV16+ Recurrent, Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate Decision
Sponsor: SQZ Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COMMANDER-001
Record Dates: First submitted 2022-04-18; First posted 2022-05-03 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Adult Solid Tumor
Keywords: recurrent cancer; metastatic; locally advanced; cancer; head and neck cancer; cervical; anal; vulvar; penile; SQZ-eAPC-HPV; HPV16; human papillomavirus 16; eAPC; enhanced antigen presenting cells; cell therapy; pembrolizumab; checkpoint inhibitors; immunotherapy; solid tumor; therapeutic vaccine; advanced solid tumor; throat cancer
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Neoplasms; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A Monotherapy Dose Escalation Phase (Experimental): In Part 1A, SQZ-eAPC-HPV as a monotherapy is administered every 3 weeks for up to a year.
  There are 3 groups ("Cohorts") in this Phase as follows:
  * Cohort 1: low dose SQZ-eAPC-HPV
  * Cohort 2: intermediate dose SQZ-eAPC-HPV
  * Cohort 3: high dose SQZ-eAPC-HPV
  Additional provisional cohorts may be opened prior to starting Part 1B.
  Interventions: Biological: SQZ-eAPC-HPV
- Part 1B Combination Phase (Experimental): In Part 1B, SQZ-eAPC-HPV is administered in combination with immune checkpoint inhibitor pembrolizumab. SQZ-eAPC-HPV will be administered on Day 1 of Cycle 1 and 200 mg of pembrolizumab will be administered on Day 8 of Cycle 1. In future cycles, patients will be first administered SQZ-eAPC-HPV and then pembrolizumab on the first day of each cycle, every 3 weeks for a maximum of 1 year for SQZ-eAPC-HPV, and 2 years for pembrolizumab.
  Interventions: Biological: SQZ-eAPC-HPV; Biological: Pembrolizumab
- Part 2 Lead-in Combination Phase (Experimental): In Part 2, SQZ-eAPC-HPV will be administered on Day 1 of each treatment cycle. Treatment with 200 mg of pembrolizumab will begin in Cycle 3. Starting at Cycle 3, patients will be administered SQZ-eAPC-HPV and then pembrolizumab every 3 weeks for a maximum of 1 year for SQZ-eAPC-HPV, and 2 years for pembrolizumab.
  Interventions: Biological: SQZ-eAPC-HPV; Biological: Pembrolizumab

INTERVENTIONS:
Biological: SQZ-eAPC-HPV — Enhanced antigen presenting cells (eAPC) cell therapy; therapeutic vaccine engineered from autologous peripheral blood mononuclear cells (PBMCs) by incorporating 5 mRNAs.
Biological: Pembrolizumab — programmed cell death 1 (PD-1) blocking antibody
  Arms: Part 1B Combination Phase; Part 2 Lead-in Combination Phase

SUMMARY:
This is a Phase 1/2, first-in-human, open label, multicenter study to assess safety and tolerability, antitumor activity, and immunogenic and pharmacodynamic effects of SQZ-eAPC-HPV as monotherapy and in combination with pembrolizumab in patients with recurrent, locally advanced, or metastatic HPV16+ solid tumors. The study includes patients with head and neck, cervical, anal, vulvar, or penile cancer.

ELIGIBILITY:
Inclusion Criteria - All Patients:

* Male or female patients ≥18 years of age
* Histologically confirmed incurable or metastatic solid tumors that are HPV16+ (performed during screening locally or centrally, or based on documented historic test results)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1
* At least 1 measurable lesion according to RECIST 1.1
* Must have a lesion that can be biopsied with acceptable clinical risk and agree to have a fresh biopsy at Screening and on Cycle 2 Day 8 (+/- 2 days)
* Patients must agree to venous access for leukapheresis and be willing to have a central line inserted if venous access is an issue
* Adequate organ function and bone marrow reserve performed within 14 days prior to leukapheresis

Inclusion Criteria - Part 2:

• Patients must not have been treated with immune check-point inhibitors

Exclusion Criteria - All Patients:

* Treatment with anticancer therapy, including investigational therapy, within 2 weeks prior to leukapheresis.
* Systemic treatment with either corticosteroids (>10 mg of prednisone or the equivalent per day) or other immunosuppressive medications within 14 days prior to leukapheresis
* Patients treated with non-corticosteroid based immunosuppressive agents within the last 6 months prior to leukapheresis
* Patients with active, known, or suspected autoimmune disease may not be eligible and should be discussed with the Sponsor
* Patients with >Grade 1 AEs related to previous treatment with anticancer or investigational therapy that do not resolve at least 2 weeks prior to leukapheresis, except Grade 2 neuropathy, ototoxicity, mucositis, fatigue, alopecia, or endocrine disorders managed with hormone replacement
* Known HIV infection, active hepatitis B or hepatitis C, or active mycobacterium tuberculosis infection
* Has known active central nervous system metastases
* Have active interstitial lung disease and any history of myocarditis
* Major surgery within 2 weeks of leukapheresis

Exclusion Criteria - Part 1B:

* Known hypersensitivity to pembrolizumab
* History of any Grade 3 immune-related AE (irAE) from prior immunotherapy

Exclusion Criteria - Part 2:

• Prior treatment with an immune check-point inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs; all, related, serious, and of special interest) as assessed by CTCAE version 5.0 | Through 6 weeks after the patient's last dose of investigational product
  For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Number of participants with dose-limiting toxicity (DLT) | Through Day 28
  For SQZ-eAPC-HPV as a monotherapy (Part 1A).
Number of participants with dose-limiting toxicity (DLT) | Through Day 42
  For SQZ-eAPC-HPV in combination with pembrolizumab (Part 1B).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of complete response [CR] and/or partial response [PR] as defined by RECIST v1.1 criteria. For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Best overall response (BoR) | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product
  Evaluation of the BoR defined as CR, PR, Stable Disease [SD], Progressive Disease [PD] or Not Evaluable [NE] as defined by RECIST v1.1 criteria. For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Progression-free survival (PFS) | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Defined as the time from first dose of study treatment to first overall response of PD by RECIST v 1.1 or to death by any cause. This will be censored at the last RECIST v1.1 assessment if PD/death is not observed. For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Duration of Response (DoR) | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Defined as the time from overall response of CR or PR to first overall response of PD by RECIST v1.1 or to death by any cause. This is defined only for patients who have a CR or PR and will be censored at the last RECIST v1.1 assessment if PD/Death is not observed. For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Disease-control rate (DCR) | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of CR or PR or SD as defined by RECIST v1.1 criteria. For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Overall survival (OS) | Through study completion, up to 2 years
  Defined as the time from first dose of study treatment to death by any cause. This will be censored at the last date patient is known to be alive if death is not observed. For SQZ-eAPC-HPV as a monotherapy, in combination with pembrolizumab, and as a monotherapy lead-in with pembrolizumab (Part 1A, Part 1B, and Part 2, respectively).
Amount of investigational product (IP) from individual patient blood collection - batch yield | From leukapheresis through manufacture, a maximum of 28 days
  To determine manufacturing feasibility as assessed by batch yield (number of manufacturing runs)
Amount of investigational product (IP) from individual patient blood collection - product failures | From leukapheresis through manufacture, a maximum of 28 days
  To determine manufacturing feasibility as assessed by number of product failures

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - University of Colorado Anschutz Cancer Pavillion, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee